CLINICAL TRIAL: NCT04118855
Title: Phase II Study of Toripalimab Combined With Axitinib as Neoadjuvant Therapy in Patients With Non-metastatic Locally Advanced Nonmetastatic Clear Cell Renal Cell Carcinoma
Brief Title: Toripalimab Combined With Axitinib as Neoadjuvant Therapy in Patients With Non-metastatic Locally Advanced Nonmetastatic Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo-RCC
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Neoadjuvant Therapy of Non-metastatic Locally Advanced Renal Cell Carcinoma
Keywords: neoadjuvant therapy; Toripalimab; axitinib; nephrectomy; partial nephrectomy
MeSH Terms: interventions — toripalimab; spartalizumab; Axitinib

STUDY DESIGN:
Intervention Model Description: Before surgery, patients will receive axitinib 5 mg bid combined with Toripalimab 3mg/KG q3w for up to 12 wk.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant arm (Experimental): Patients will receive axitinib 5 mg bid combined with Toripalimab 3mg/KG q3w for up to 12 wk.
  Interventions: Drug: Toripalimab; Drug: Axitinib

INTERVENTIONS:
Drug: Toripalimab — 240mg, IV (in the vein) on on day 1 of 3-week, 6-week and 9-week for a total of 3 doses prior to partial nephrectomy or radical nephrectomy
  Other Names: anti-PD-1 monoclonal antibody
Drug: Axitinib — 5 mg by mouth twice each day for 12 weeks prior to nephrectomy

SUMMARY:
This study is design to prospectively investigate the safety and efficacy of Toripalimab combined with Axitinib in downsizing tumors in patients with nonmetastatic biopsy-proven clear cell renal cell carcinoma. Toripalimab is new antibody that may help activate the immune system by blocking the function of an inhibitory molecule, Programmed cell death-1 (PD-1). This is a single-institution, single-arm phase 2 clinical trial.

DETAILED DESCRIPTION:
This study is design to prospectively investigate the safety and efficacy of Toripalimab combined with Axitinib in downsizing tumors in patients with nonmetastatic biopsy-proven clear cell renal cell carcinoma. Toripalimab is new antibody that may help activate the immune system by blocking the function of an inhibitory molecule, Programmed cell death-1 (PD-1). This is a single-institution, single-arm phase 2 clinical trial. Patients will receive axitinib 5 mg bid combined with Toripalimab 3mg/KG q3w for up to 12 wk. Patients then will receive partial or radical nephrectomy after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic biopsy-proven clear cell renal cell carcinoma (T2-T3N0-1M0)
* Schedule to undergo either partial or radical nephrectomy as part of treatment plan
* ECOG performance status of 0 or 1
* Adequate organ and marrow function defined by study-specified laboratory tests
* Agree to comply with scheduled visits, treatment plans, lab tests and other study procedures
* Do not have any other cancers in the 5 yr preceding diagnosis of their renal cancer

Exclusion Criteria:

* Patients who have received other systems for anti-tumor treatment
* Patients who have previously received targeted or immunotherapy
* Need for urgent or emergent nephrectomy to relieve symptoms
* Current use of immunosuppressive agents
* Pregnant or breastfeeding women
* History of autoimmune disease or syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Objective Tumor Response Rate | 3 month
  Number of patients achieving a complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors

SECONDARY OUTCOMES:
Safety assessed by adverse events | through study completion, an average of 4 months
  Safety as assessed by number of participants experiencing adverse events
Perioperative complication rate | from perioperative to 90 days after surgery
  Perioperativecomplications judged by Clavien-Dindo classification
Quality of Life questionnaire | Baseline, 3 weeks, 12 weeks and after surgery
  Quality of Life as assessed by the Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI) -15 questionnaire
Tumor complexity changing by total R.E.N.A.L. score | Baseline, 12 weeks
  R.E.N.A.L. Nephrometry Score) to quantify the anatomical characteristics of renal R.E.N.A.L. score consists of 5 anatomical features, and sum them up.

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

REFERENCES:
- [Derived] Huang J, Wang Y, Xu F, Wang Z, Wu G, Kong W, Cheoklong NG, Tricard T, Wu X, Zhai W, Zhang W, Zhang J, Zhang D, Chen S, Lian Y, Chen Y, Zhang J, Huang Y, Xue W. Neoadjuvant toripalimab combined with axitinib in patients with locally advanced clear cell renal cell carcinoma: a single-arm, phase II trial. J Immunother Cancer. 2024 Jun 11;12(6):e008475. doi: 10.1136/jitc-2023-008475. PMID 38862251